CLINICAL TRIAL: NCT03346707
Title: 10.5T Safety and Feasibility Study
Brief Title: Safety and Feasibility of Imaging at 10.5 Tesla
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: RAD-2017-24570
Record Dates: First submitted 2017-09-22; First posted 2017-11-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- 10.5 Tesla
  Interventions: Device: 10.5 Tesla

INTERVENTIONS:
Device: 10.5 Tesla — 10.5Tesla MR scan

SUMMARY:
This unique NMR instrument is the first of its kind, and the most advanced system that is capable of brain, torso and extremity imaging in humans at such a high magnetic field. It will be transformative in performance relative to 7Tesla, and significantly expand the capabilities of multinuclear MRI, fMRI, morphological imaging, MRS etc. in the human brain and body.

In addition, to the known and potential benefits of performing anatomic and functional imaging studies at 10.5T, there are also known short-term side effects associated with subjecting humans to such high magnetic fields. This protocol will study the magnitude and variability of the short term and long term physiological, cognitive and vestibular effects while also assessing the feasibility of acquiring the types of data needed for translating research protocols onto this higher field strength scanner.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 70
2. Able to self-consent
3. Weight less than 190 pounds
4. Participated in high field MRI studies (7T or higher)

Exclusion Criteria:

Subjects with metallic, magnetic, and/or electrically conductive implants or external devices.

1. Ferromagnetic implants
2. Any foreign metal objects in the body
3. History of shrapnel or shot gun injury
4. Cardiac pacemakers
5. Defibrillator
6. Neuronal stimulator
7. Magnetic aneurysm clip
8. Large tattoos on the abdomen or the brain and neck
9. Hip replacement
10. Too large to fit in the magnet (body mass index >= 40, approx.)
11. Severe claustrophobia
12. Women who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controsl
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Physiologic effects of human exposure to 10.5T (Blood Pressure). | Baseline and 2-4 weeks
  Change in blood pressure will be studied when exposed to 10.5T. Systolic and diastolic pressures (mmHg) will be measured before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Physiologic effects of human exposure to 10.5T (Heart Rate). | Baseline and 2-4 weeks
  Change in heart rate will be studied when exposed to 10.5T. Heart rate (beats per minute) will be measured before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Physiologic effects of human exposure to 10.5T (Peripheral Capillary Oxygen Saturation (SPO2)). | Baseline and 2-4 weeks
  Change in peripheral capillary oxygen saturation will be studied when exposed to 10.5T. Peripheral capillary oxygen saturation (%) will be measured before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Physiologic effects of human exposure to 10.5T (Respiration Rate). | Baseline and 2-4 weeks
  Change in respiration rate will be studied when exposed to 10.5T. Respiration rate (breaths per minute) will be measured before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Cognitive effects of human exposure to 10.5T (Brief Fatigue Inventory). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Brief Fatigue Inventory. Brief Fatigue Inventory (average score) will be administered before first 10.5T exposure, day after first 10.5T exposure, before second 10.5T exposure, and day after second 10.5T exposure.
Cognitive effects of human exposure to 10.5T (Letter Number Sequencing). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Letter Number Sequencing. Letter Number Sequencing (total raw score) will be administered before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Cognitive effects of human exposure to 10.5T (Digit Span Test). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Digit Span Test. Digit Span Test (total raw score) will be administered before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Cognitive effects of human exposure to 10.5T (Hopkins Verbal Test). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Hopkins Verbal Test. Hopkins Verbal Test (total recall, delayed recall, retention %, recognition discrimination index) will be administered before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Cognitive effects of human exposure to 10.5T (Symbol Digit Modalities Test). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Symbol Digit Modalities Test. Symbol Digit Modalities Test (# correct in 90 seconds) will be administered before first 10.5T exposure after first 10.5T exposure, before second 10.5T exposure, and after second 10.5T exposure.
Cognitive effects of human exposure to 10.5T (Trail Making Test). | Baseline and 2-4 weeks
  Change in cognitive function will be studied when exposed to 10.5T using Trail Making Test. Trail Making Test (time to completion) will be administered before first 10.5T exposure after first 10.5T exposure, before second 10.5T exposure, and after second 10.5T exposure.
Vestibular effects of human exposure to 10.5T (Activity-specific Balance Confidence Scale). | Baseline and 2-4 weeks
  Change in vestibular function will be studied when exposed to 10.5T using Activity-specific Balance Confidence Scale. Activity-specific Balance Confidence Scale (% of self confidence) will be administered before first 10.5T exposure, day after first 10.5T exposure, before second 10.5T exposure, and day after second 10.5T exposure.
Vestibular effects of human exposure to 10.5T (Smooth Pursuit). | Baseline and 2-4 weeks
  Change in vestibular function will be studied when exposed to 10.5T using smooth pursuit test. Smooth pursuit test (# of saccades for 4 types of eye movements) will be administered before, during, and after 10.5T exposure at baseline and 2-4 weeks later.
Vestibular effects of human exposure to 10.5T (Spontaneous Eye Movement). | Baseline and 2-4 weeks
  Change in vestibular function will be studied when exposed to 10.5T using spontaneous eye movement test. Spontaneous eye movement test (# of saccades with and without fixation) will be administered before, during, and after 10.5T exposure at baseline and 2-4 weeks later.

CONTACTS AND LOCATIONS:
Locations (1):
- CMMR, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No